CLINICAL TRIAL: NCT06960733
Title: Comparative Efficacy of Winged Versus Traditional Plastic Stents for Biliary Drainage in Benign and Malignant Obstructions: A Randomized Study
Brief Title: Comparison Between Winged Versus Traditional Plastic Stents for Biliary Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Viaduct-ERCP
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2010-10

CONDITIONS: Biliary Obstruction; Bile Duct Stones; Biliary Tract Cancer
Keywords: ERCP; Biliary obstruction; biliary stenting; plastic stent
MeSH Terms: conditions — Cholecystolithiasis; Biliary Tract Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Stenting (Active Comparator): Stenting of biliary tract by standard plastic stent. Change of stent-type at regular stent exchange after three months (from winged to standard and vice versae).
  Interventions: Device: Winged plastic stent; Device: Standard plastic stents
- Winged Stent (Experimental): Stenting of biliary tract by use of winged-design stent. Change of stent-type at regular stent exchange after three months (from winged to standard and vice versae).
  Interventions: Device: Winged plastic stent; Device: Standard plastic stents

INTERVENTIONS:
Device: Winged plastic stent — Patient with need for stenting of bile duct were randomised for kind of stents. Stents used were either standard plastic stents or stents with winged design. In this Intervention winged stents were used.
Device: Standard plastic stents — Patient with need for stenting of bile duct were randomised for kind of stents. Stents used were either standard plastic stents or stents with winged design. In this Intervention standard plastic stents were used.

SUMMARY:
This study was randomized, controlled, blinded trial with a two-arm parallel-group design to directly compare the therapeutic outcomes of winged versus conventional stents in patients with benign or malignant biliopancreatic conditions requiring ERCP and subsequent insertion or replacement of plastic stents.

DETAILED DESCRIPTION:
Procedure The study was structured as a randomized, controlled trial using a two-arm parallel group design to compare different therapies (winged stent vs. conventional stent). Randomization was carried out in a 1:1 ratio using block randomization. Upon stent exchange, participants were switched to the alternate treatment group. Each subject was intended to receive both forms of therapy over the course of the treatment periods in a crossover design, with only the sequence of therapies being determined randomly (Figure 1).

The procedures were conducted using standard techniques. No additional steps, biopsies, or similar procedures were required. For the ERCPs carried out in the Endoscopy Department of the University Hospital Leipzig, Fujifilm video duodenoscopes were utilized

Data On the procedure date, we gathered essential baseline and procedural information including demographic data (age and gender), previous stent interventions, diagnostic imaging and laboratory results, specifics of the stent used (type, diameter, and length), the effectiveness of the stent insertion, and any associated complications.

Beyond standard care, follow-up was conducted at intervals of one week, one month, and two months post-intervention, utilizing a methodical questionnaire to monitor clinical progress and evaluate for any stent-related dysfunction."

ELIGIBILITY:
Inclusion Criteria:

* Biliopancreatic disorder requiring plaxtic biliary stent therapy
* written informed consent

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Live Expectancy of less than one month
* Biliary drainage by metal stent or external drainage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2013-04-30 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Dysfunction | 3 Months
  Sign of dysfunction of biliary stenting (fever, pain, jaundice)

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Hoffmeister, Professor, Study Chair — University of Leipzig Medical Center
Locations (1):
- University of Leipzig Medical Center, Department of Gastroenterology, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No